CLINICAL TRIAL: NCT02025673
Title: Study of Betatrophin Levels in Patients With Type 2 Diabetes and Gestational Diabetes and Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Jing Dong, associate professor, Qingdao University
Other Study IDs: Betatrophin-Human
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Pregnancy; Gestational Diabetes Mellitus (GDM); Type 2 Diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy Controls: Healthy subjects as control group.
- Type 2 diabetes: Patients with type 2 diabetes.
- Gestational diabetes mellitus: Patients with gestational diabetes mellitus.

SUMMARY:
Betatrophin is a newly identified hormone that promotes pancreatic beta cell proliferation, improves glucose tolerance and regulates lipids metabolism. A recent study showed that circulating concentrations of betatrophin doubled in type 1 diabetes. The objective of this study is to investigate the association of serum betatrophin levels with the progression of diabetic retinopathy in patients with type 2 diabetes and the level of betatrophin in gestational diabetes patients and pregnant women.

DETAILED DESCRIPTION:
200 subjects were recruited in this study and divided into six groups for comparison of the serum betatrophin. 70 healthy subjects and 20 healthy young volunteers were enrolled for investigating the role of betatrophin in energy homeostasis and the circadian rhythm. 50 patients with type 2 diabetes were classified into three groups by the stage of diabetic retinopathy. Rank test was used to analyze the correlation between the progression of diabetic retinopathy and circulating betatrophin. Betatrophin were measured by a commercially available enzyme-linked immunosorbent assay and confirmed via Western Blot.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients
* Patients with HbA1c >or= 7.0%

Exclusion Criteria:

* Participation in other investigational Clinical Trial
* Type 1 diabetes mellitus patients
* Patients with history of severe hepatic dysfunction
* Treatment with antifungal agent especially Miconazole
* Patients with active smoking or history of smoking cessation less than 2 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 19 healthy pregnant women and 9 pregnant women with gestational diabetes mellitus (GDM) were enrolled in the study. 24 patients with newly diagnosed type 2 diabetes mellitus before treatment, 35 patients with type 2 diabetes mellitus after treatment. Subjects were recruited from patients at the Department of Clinical Endocrinology and Maternity Department, Affiliated Hospital of Qingdao University.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Serum levels of betatrophin in type 2 diabetes patients, gestational diabetes patients and pregnant women | Up to one month

SECONDARY OUTCOMES:
Correlation of betatrophin concentration with other variables | Up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Jing Dong, Ph.D, Principal Investigator — Medical College of Qingdao University

REFERENCES:
- [Result] Espes D, Lau J, Carlsson PO. Increased circulating levels of betatrophin in individuals with long-standing type 1 diabetes. Diabetologia. 2014 Jan;57(1):50-3. doi: 10.1007/s00125-013-3071-1. PMID 24078058